CLINICAL TRIAL: NCT01976598
Title: Sub-Sensory Intraspinal Neurostimulation Therapy In the Treatment of Neuropathic Back and/or Leg Pain
Brief Title: Sub-Sensory Intraspinal Neurostimulation Therapy
Status: Terminated | Type: Observational
Why Stopped: Protocol proved too cumbersome. Consequently, only one one patient enrolled, and completed.
Sponsor: Algos Clinical Development Thomas L. Yearwood, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Algos Clinical Development Thomas L. Yearwood, MD, PhD, Medical Director / Principal Investigator, Algos Clinical Development
Organization: Algos Clinical Development (Other)
Other Study IDs: ALG-ANA1001; 20131546 (Other: Western Institutional Review Board (WIRB®))
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Back Pain; Back Pain With Radiation; Pain in Leg, Unspecified
Keywords: chronic; back; leg; pain; sub-sensory; stimulation; Neuromodulation; Yearwood
MeSH Terms: conditions — Back Pain; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Cord Stimulation: Sub-Sensory: Patients implanted with a Boston Scientific Spinal Cord Stimulation System for the treatment of chronic back and/or leg pain using Sub-Sensory Stimulation.
  Interventions: Other: Sub-Sensory Stimulation

INTERVENTIONS:
Other: Sub-Sensory Stimulation — Sub-Sensory Stimulation using Boston Scientific Spinal Cord Stimulation System in patients currently implanted with the system .
  Other Names: Sub-Sensory Spinal Cord Stimulatiocn.

SUMMARY:
To explore the optimal stimulation parameters and locations for sub-perception programming in patients with previously implanted spinal cord stimulation systems for the treatment of chronic back and/or leg pain.

DETAILED DESCRIPTION:
Chronic pain remains a serious public health problem, resulting in approximately 100 million chronic pain patients in the U.S. alone [1]. While numerous treatments exist, none completely addresses this issue. In particular, spinal cord stimulation (SCS) has become an established technique for treating patients with chronic neuropathic pain [2]. The conventional paradigm for SCS treatment is to attempt to mask the pain by substituting the pain sensation with paresthesias [3]; however, newer studies have shown that it is possible to gain excellent pain relief without concomitant paresthesias ("sub-threshold stimulation") using different stimulation parameters [4] [5]. Because these paresthesia-free programming paradigms are still new, the best to place the stimulation and the best programming parameters to use is still unclear, making it difficult to place the leads during surgical implantation and to program the patient afterwards. Additionally, sub-threshold stimulation does not provide immediate pain relief, but may take several hours or even days to feel relief, making a simple programming session of a few hours insufficient to determine the optimal stimulation placement. While these differences from conventional SCS make programming more difficult initially, studying this new stimulation paradigm, especially differences in optimal stimulation location and the time course of pain relief, may also provide insight into the mechanism of action of sub-threshold stimulation. This protocol aims to study the optimal stimulation parameters and locations with SCS using sub-threshold stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary pain complaint of persistent or recurrent low back and/or leg pain, with or without leg pain, for at least 180 days prior to Baseline.
* Received a Boston Scientific SCS System with active contacts located between superior endplate of T7 and the inferior endplate of T10 with a minimum of three active contacts within this anatomical area.
* No back surgery within 180 days prior to Baseline.
* Has had stimulator "on" (activated or operational) for at least 36 hours prior to Baseline evaluation.
* Average low back and/or leg pain intensity, during the position/activity which routinely causes worst pain, of 5 or greater on a 0-10 numerical rating scale without neurostimulation.
* If taking prescription opioids for primary chronic pain complaint (low back and/or leg pain), must have been on a stable prescription (same drug(s) and dose(s)) for 30 days prior to Baseline
* Consumed an average total daily morphine equivalent of ≤300 mg during the 30 days prior to Baseline
* Willing and able to comply with all protocol-required procedures and assessments/evaluations (e.g. willing to comply with opioid prescription lock throughout the study, changes to the stimulation parameters, complete twice-daily diary)
* 22 years of age or older when written informed consent is obtained
* Able to independently read and complete all questionnaires and assessments provided in English
* Subject signed a valid, IRB-approved informed consent form (ICF) provided in English

Exclusion Criteria:

* Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment, might confound reporting of study outcomes (e.g. pelvic pain, chronic migraine, schizophrenia)
* Current uncontrolled diabetes mellitus
* Significant cognitive impairment at Baseline that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to assess pain intensity and/or complete a pain diary
* Participated in any investigational study within 30 days prior to the Screening Visit or is currently participating in another clinical trial that may influence the data that will be collected for this study
* A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception
* Plan to receive any massage or manipulation directly over the leads or by the location of the IPG or treatments that involve sudden jerking motions of the torso at any time during the course of the study
* Unresolved active litigation related to the pain condition being treated in the study
* Currently involved in a worker's compensation claim
* Unable to operate the SCS System

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a Boston Scientific Spinal Cord Stimulation System for the treatment of chronic back and/or leg pain
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score (VAS) | 32 days
  The primary outcome measure is the final visual analog score (VAS) score obtained using a paper pain diary obtained on the last evening of each program.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Yearwood, MD, PhD, Principal Investigator — Algos Cinical Development
Locations (1):
- Comprehensive Pain and Rehabilitation, Pascagoula, Mississippi, United States

REFERENCES:
- [Background] Tiede J, Brown L, Gekht G, Vallejo R, Yearwood T, Morgan D. Novel spinal cord stimulation parameters in patients with predominant back pain. Neuromodulation. 2013 Jul-Aug;16(4):370-5. doi: 10.1111/ner.12032. Epub 2013 Feb 21. PMID 23433237
- See also: Home Page for the Food and Drug Administration (FDA) — http://www.fda.gov
- See also: WIRB sets the standard in the field of independent ethical review of biomedical research on human subjects. — http://www.wirb.com